CLINICAL TRIAL: NCT01354314
Title: Pilot Study of Paroxetine and Fluconazole for the Treatment of HIV Associated Neurocognitive Disorder (HAND)
Brief Title: Study of Paroxetine and Fluconazole for the Treatment of HIV Associated Neurocognitive Disorder
Acronym: ParaFlu
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ned Sacktor, Professor of Neurology, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00037283; P30MH075673-05 (NIH)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: HIV Associated Neurocognitive Disorder
Keywords: HIV; Neurocognitive impairment; Memory; Dementia; CSF marker; Functional assessment; MRS; Magnetic resonance spectroscopy; Arterial spin labeling; SSRI
MeSH Terms: conditions — Dementia | interventions — Fluconazole; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fluconazole (Experimental): Fluconazole 100 mg every 12 hours orally per day; placebo in place of paroxetine
  Interventions: Drug: Fluconazole
- Paroxetine (Experimental): Paroxetine 20 mg orally once per day; placebo in place of fluconazole
  Interventions: Drug: Paroxetine
- Paroxetine and Fluconazole (Experimental): Fluconazole 100 mg every 12 hours orally per day and paroxetine 20 mg every evening orally per day
  Interventions: Drug: Paroxetine and Fluconazole
- Placebo (Placebo Comparator): Placebo in place of both fluconazole and paroxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluconazole — One 100 MG capsule taken twice daily, 12 hour dosing
  Arms: Fluconazole
Drug: Paroxetine — Two 10 MG capsules paroxetine once daily in the evening
  Arms: Paroxetine
Drug: Paroxetine and Fluconazole — One capsule 100 MG fluconazole every 12 hours orally per day; Two 10 MG capsules paroxetine orally once daily in the evening
  Arms: Paroxetine and Fluconazole
Drug: Placebo — One capsule in the morning, three capsules in the evening
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if paroxetine and fluconazole are safe and effective as a treatment for problems with memory, concentration, thinking, and judgment in people who are infected with HIV. Paroxetine is an antidepressant approved by the FDA to treat major depression. Fluconazole is an antifungal medication approved by the FDA to treat fungal infections.

DETAILED DESCRIPTION:
The study will be a 24 week double-blind, placebo-controlled 2x2 factorial design pilot Phase I/II study in 60 HIV+ individuals with HAND. Participants will be randomly assigned to one of four groups: 1) fluconazole 100 mg every 12 hours orally per day, 2) paroxetine 20mg every evening orally per day, 3) fluconazole 100mg every 12 hours orally per day and paroxetine 20mg every evening orally per day and 4) placebo.

Primary Aim: To obtain preliminary data to evaluate the efficacy of fluconazole and/or paroxetine to decrease CSF lipid and protein markers of oxidative stress [CSF ceramide and (C18:0 levels) and 3-nitrosylated proteins].

Secondary Aims:

i) To evaluate the safety and tolerability of fluconazole and/or paroxetine in HIV+ individuals with HAND ii) To evaluate the effect of fluconazole and/or paroxetine on neurocognitive performance in HIV+ individuals with HAND iii) To evaluate the effect of fluconazole and/or paroxetine on functional performance in HIV+ individuals with HAND iv) To evaluate the CNS penetration of fluconazole and paroxetine after 24 weeks of treatment v) To obtain preliminary data to evaluate the efficacy of fluconazole and/or paroxetine to improve abnormal imaging markers as measured by magnetic resonance spectroscopy (MRS) and arterial spin labeling

ELIGIBILITY:
Inclusion Criteria:

* HIV+ based on ELISA and confirmed by either Western blot or plasma HIV RNA
* capable of providing informed consent
* age range: 18-65 years
* presence of neuropsychological testing impairment as defined by performance at least 1.0 standard deviation below age-matched and education-matched controls on three or more independent neuropsychological tests at the screening visit, or performance at least 2.0 standard deviations below age-matched and education-matched controls on one independent neuropsychological test and at least 1.0 standard deviation below age-matched and education-matched controls on a second independent neuropsychological test at the screening visit
* a stable HAART regimen for 3 months with no plans to change the antiretroviral regimen over the study period (confirmed by discussion with a patient's primary provider)
* the following lab values within 2 weeks prior to entry: hemoglobin > 8.9 g/dl, absolute neutrophil count > 500 cells/mm3, platelet count > 50,000 cells/mm3, ALT < 2.5 X upper limit of normal, alkaline phosphatase < 3 X upper limit of normal, serum creatinine >= 2 X upper limit of normal
* a negative serum or urine beta-HCG pregnancy test for all women of reproductive potential (have not reached menopause or undergone hysterectomy, oophorectomy, or tubal ligation)
* neurological examination by a physician revealing no contraindication to a lumbar puncture. If an examination suggests a possible space-occupying brain mass lesion, neuroimaging with CT or MRI must confirm the absence of a mass lesion.

Exclusion Criteria:

* current or past opportunistic CNS infection (fungal or non-fungal) at study entry
* current systemic fungal infection
* current or past use of fluconazole within 30 days of the screening visit
* history or current clinical evidence of schizophrenia
* history of chronic neurological disorder such as multiple sclerosis or uncontrolled epilepsy
* active symptomatic AIDS defining opportunistic infection within 30 days prior to study entry
* history of abnormal medical illness or current severe affective disorder (e.g., depression with suicidal intention) which in the opinion of the investigators would constitute a safety risk for patients or interfere with the ability of a patient to complete the study
* treatment with anticoagulants including coumadin, heparin, or low molecular weight heparin which would be a contraindication for the lumbar puncture
* HIV+ individuals with moderate or severe confounding illnesses
* prior use of SSRI's within 1 month of screening
* active substance abuse (illicit drugs and/or controlled medications) or active severe alcohol abuse, evidenced by history intake or urine toxicology at any visit prior to study entry (starting study medication)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Sacktor, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Institute for Clinical and Translational Research, Adult Outpatient Clinical Research Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxetine: Paroxetine 20 mg orally once per day; placebo in place of fluconazole every 12 hours orally per day
  Paroxetine: Two 10 MG capsules paroxetine once daily in the evening
- Fluconazole: Fluconazole 100 mg every 12 hours orally per day; placebo in place of paroxetine every evening orally per day
  Fluconazole: One 100 MG capsule taken twice daily, 12 hour dosing
- Placebo: Placebos in place of fluconazole and paroxetine
  Placebos: One capsule placebo #1 every 12 hours orally per day; Two capsules placebo #2 orally once daily in the evening
Period: Overall Study
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Started | 12 | 11 | 11 | 11
Completed (ITT) (Completed trial with evaluable data for intention to treat analysis.) | 11 | 11 | 9 | 10
Completed (Per protocol: evaluable outcome measures and 90+ percent of target study treatment total dose.) | 6 | 8 | 3 | 5
Not Completed | 6 | 3 | 8 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Less than 90% Adherence | 4 | 2 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.83 (5.77) | 52.00 (6.62) | 51.73 (5.76) | 48.73 (10.23) | 50.56 (7.17)
Age, Customized [Number; unit: Years]
  25 to 34 | 0 | 0 | 0 | 1 | 1
  35 to 44 | 2 | 1 | 1 | 1 | 5
  45 to 54 | 8 | 7 | 7 | 5 | 27
  55 to 64 | 2 | 3 | 3 | 4 | 12
Sex/Gender, Customized [Number; unit: participants]
  Male | 4 | 9 | 10 | 9 | 32
  Female | 7 | 2 | 1 | 1 | 11
  Transgender (Male to Female) | 1 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 11 | 11 | 11 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 8 | 10 | 9 | 37
  White | 2 | 3 | 1 | 1 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Education [Mean (Standard Deviation); unit: Years Completed] | 11.83 (2.08) | 12.36 (1.80) | 12.91 (1.87) | 12.36 (2.11) | 12.36 (1.94)
Years Since HIV Diagnosis [Mean (Standard Deviation); unit: Years] — Based on self-report from participants.
  Years | 15.33 (6.77) | 16.36 (7.90) | 15.45 (6.76) | 17.36 (7.93) | 16.11 (7.14)
Absolute CD4 Count [Mean (Standard Deviation); unit: Cells per cubic mm] | 516.1 (244.8) | 637.3 (241.7) | 555.2 (282.8) | 510.4 (235.1) | 553.9 (248.2)
Plasma HIV Viral Load [Number; unit: participants]
  Undetectable (<50 copies/mL) | 7 | 9 | 11 | 10 | 37
  Detectable: 50-99 copies/mL | 3 | 0 | 0 | 1 | 4
  Detectable: 100-249 copies/mL | 0 | 2 | 0 | 0 | 2
  Detectable: 250-499 copies/mL | 2 | 0 | 0 | 0 | 2
Hepatitis C Infection Status [Number; unit: participants]
  Positive History | 6 | 3 | 7 | 8 | 24
  Negative History | 6 | 8 | 4 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in CSF Ceramide Between Baseline and Week 24 (C18:0 Levels) - Intent to Treat
Description: CSF lipid and protein markers of oxidative stress: Change in CSF ceramide (C18:0 levels) between baseline and week 24 for all participants for whom baseline and follow-up CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
ng/mL | -30.78 [-68.27 to 24.71] | 4.16 [-38.76 to 47.95] | -12.17 [-56.98 to 9.81] | -30.56 [-65.78 to 59.94]
Statistical Analysis 1: Comparison: Paroxetine and Fluconazole vs Placebo; Test type: Superiority; p = 0.893, Regression, Linear
Statistical Analysis 2: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.594, Regression, Linear
Statistical Analysis 3: Comparison: Fluconazole vs Placebo; Test type: Superiority; p = 0.712, Regression, Linear

2. Primary Outcome: Change in CSF Ceramide Between Baseline and Week 24 (C18:0 Levels) - Per Protocol
Description: CSF lipid and protein markers of oxidative stress: Change in CSF ceramide (C18:0 levels) between baseline and week 24 for participants with 90% or greater study drug adherence and for whom baseline and follow-up CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: For per protocol analysis, 18 participants (out of the 22 who completed the trial with 90% or greater study drug adherence) had follow-up CSF for primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
ng/mL | -51.35 [-119.66 to 5.95] | 34.11 [-4.71 to 51.20] | -65.00 [-69.00 to -60.99] | -52.37 [-87.89 to -7.96]
Statistical Analysis 1: Comparison: Paroxetine and Fluconazole vs Placebo; Test type: Superiority; p = 0.673, Regression, Linear
Statistical Analysis 2: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.153, Regression, Linear
Statistical Analysis 3: Comparison: Fluconazole vs Placebo; Test type: Superiority; p = 0.282, Regression, Linear

3. Primary Outcome: Change in CSF 3-nitrosylated Protein Levels Between Baseline and Week 24 - Intent to Treat
Description: CSF lipid and protein markers of oxidative stress: Change in 3-nitrosylated protein levels between baseline and week 24 for all participants for whom CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: For intention to treat analysis, 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: pi*mm^2
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
pi*mm^2 | 6.392 [-14.214 to 11.674] | 12.235 [-23.502 to 30.271] | 33.767 [-10.912 to 35.853] | -8.747 [-21.055 to 4.282]
Statistical Analysis 1: Comparison: Paroxetine and Fluconazole vs Placebo; Test type: Superiority; p = 0.327, Regression, Linear
Statistical Analysis 2: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.178, Regression, Linear
Statistical Analysis 3: Comparison: Fluconazole vs Placebo; Test type: Superiority; p = 0.480, Regression, Linear

4. Primary Outcome: Change in CSF 3-nitrosylated Protein Levels Between Baseline and Week 24 - Per Protocol
Description: CSF lipid and protein markers of oxidative stress: Change in 3-nitrosylated protein levels between baseline and week 24 for participants with 90% or greater adherence to study drug and for whom CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: For per protocol analysis, 18 participants (out of the total 22 who completed the trial with 90% or greater study drug adherence) had follow-up CSF for primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: pi*mm^2
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
pi*mm^2 | 0.712 [-17.441 to 10.034] | 0.257 [-31.676 to 25.563] | -3.959 [-22.821 to 14.904] | -13.160 [-19.314 to -4.499]
Statistical Analysis 1: Comparison: Paroxetine and Fluconazole vs Placebo; Test type: Superiority; p = 0.267, Regression, Linear
Statistical Analysis 2: Comparison: Paroxetine vs Placebo; Test type: Superiority; p = 0.368, Regression, Linear
Statistical Analysis 3: Comparison: Fluconazole vs Placebo; Test type: Superiority; p = 0.672, Regression, Linear

5. Secondary Outcome: Change in CSF sCD14 Between Baseline and Week 24 - Intent to Treat
Description: CSF immune and neuronal injury markers: Change in CSF sCD14 between baseline and week 24 for all participants for whom baseline and follow-up CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
pg/mL | -17.7 [-53.7 to 32.4] | 15.2 [-19.1 to 72.3] | -16.5 [-48.5 to -6.1] | 12.0 [-53.6 to 21.0]

6. Secondary Outcome: Change in CSF sCD14 Between Baseline and Week 24 - Per Protocol
Description: CSF immune and neuronal injury markers: Change in CSF sCD14 between baseline and week 24 for participants with 90% or greater study drug adherence and for whom baseline and follow-up CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
pg/mL | -4.3 [-62.0 to 60.3] | 33.2 [-55.1 to 84.7] | -5.1 [-5.6 to -4.5] | -18.9 [-51.8 to 12.0]

7. Secondary Outcome: Change in CSF CD163 Between Baseline and Week 24 - Intent to Treat
Description: CSF immune and neuronal injury markers: Change in CSF CD163 between baseline and week 24 for all participants for whom baseline and follow-up CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
ng/mL | 1.6 [-3.2 to 3.5] | -0.7 [-2.4 to 1.1] | -2.7 [-8.1 to 2.6] | -3.8 [-5.1 to 1.4]

8. Secondary Outcome: Change in CSF CD163 Between Baseline and Week 24 - Per Protocol
Description: CSF immune and neuronal injury markers: Change in CSF CD163 between baseline and week 24 for participants with 90% or greater study drug adherence and for whom baseline and follow-up CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
ng/mL | -3.2 [-6.1 to -0.2] | -0.7 [-2.5 to 3.9] | -7.5 [-9.8 to -5.1] | -1.8 [-3.8 to 0.7]

9. Secondary Outcome: Change in CSF Neurofilament Protein Light Chain (NFL) Between Baseline and Week 24 - Intent to Treat
Description: CSF immune and neuronal injury markers: Change in CSF neurofilament protein light chain (NFL) between baseline and week 24 for all participants for whom baseline and follow-up CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
pg/mL | 0.0890 [0.0285 to 0.1855] | 0.1710 [0.1043 to 0.2733] | 0.2030 [-0.0270 to 0.2170] | 0.1000 [-0.0475 to 0.1705]

10. Secondary Outcome: Change in CSF Neurofilament Protein Light Chain (NFL) Between Baseline and Week 24 - Per Protocol
Description: CSF immune and neuronal injury markers: Change in CSF neurofilament protein light chain (NFL) between baseline and week 24 for participants with 90% or greater study drug adherence and for whom baseline and follow-up CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
pg/mL | 0.0560 [0.0233 to 0.1180] | 0.1580 [-0.0012 to 0.2588] | 0.0985 [0.0358 to 0.1613] | 0.1375 [0.0528 to 0.2223]

11. Secondary Outcome: Change in CSF Neurofilament Protein Heavy Chain (pNFL) Between Baseline and Week 24 - Intent to Treat
Description: CSF immune and neuronal injury markers: Change in CSF neurofilament protein heavy chain (pNFL) between baseline and week 24 for all participants for whom baseline and follow-up CSF data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: 31 participants, out of the total 45 enrolled, completed the trial with follow-up CSF primary outcome measures.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 11 | 8 | 5 | 7
pg/mL | -0.0080 [-0.0275 to 0.0205] | 0.0705 [0.0338 to 0.0975] | 0.0400 [0.0290 to 0.1280] | 0.0520 [0.0345 to 0.0755]

12. Secondary Outcome: Change in CSF Neurofilament Protein Heavy Chain (pNFH) Between Baseline and Week 24 - Per Protocol
Description: CSF immune and neuronal injury markers: Change in CSF neurofilament protein heavy chain (pNFH) between baseline and week 24 for participants with 90% or greater study drug adherence and for whom baseline and follow-up CSF data are available (per protocol analysis).
Time Frame: 24 Weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
Number analyzed (Participants) | 6 | 6 | 2 | 4
pg/mL | -0.0035 [-0.0208 to 0.0303] | 0.0645 [0.0133 to 0.0888] | 0.0270 [0.0205 to 0.0335] | 0.0395 [0.0130 to 0.0618]

13. Secondary Outcome: Neurocognitive Performance: Trail Making A - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the Trail-making test, part A speed of completion (Z scores).
Time Frame: 24 Weeks
Population: Includes all participants who completed the study with test data available at the Baseline and Week 24 visits for Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 9 | 10 | 10
Z score | 0.045 (0.88) | 0.067 (0.98) | 0.000 (0.77) | 0.09 (0.89)

14. Secondary Outcome: Neurocognitive Performance: Trail Making A - Per Protocol
Description: as for outcome 13
Time Frame: 24 Weeks
Population: Per protocol analysis: Includes all participants who completed the study per protocol and with test data available at the Baseline and Week 24 visits.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | -0.28 (0.96) | 0.17 (0.98) | 0.24 (0.58) | 0.52 (1.01)

15. Secondary Outcome: Neurocognitive Performance: Trail Making B - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the Trail-making test, part B speed of completion (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 9 | 10 | 10
Z score | 0.47 (0.98) | -0.71 (0.93) | 0.51 (1.03) | 0.020 (0.75)

16. Secondary Outcome: Neurocognitive Performance: Trail Making B - Per Protocol
Description: as for outcome 15
Time Frame: 24 Weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | 0.63 (0.95) | -0.83 (1.48) | 0.49 (0.89) | 0.16 (0.50)

17. Secondary Outcome: Neurocognitive Performance: Grooved Pegboard, Dominant - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the Grooved Pegboard test, dominant hand speed of completion (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 8 | 10 | 10
Z score | 0.23 (0.92) | 0.05 (1.09) | 0.57 (1.05) | -0.01 (0.88)

18. Secondary Outcome: Neurocognitive Performance: Grooved Pegboard, Dominant - Per Protocol
Description: as for outcome 17
Time Frame: 24 Weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | 0.15 (1.10) | -0.67 (0.61) | 0.59 (1.23) | -0.14 (1.07)

19. Secondary Outcome: Neurocognitive Performance: Grooved Pegboard, Non-Dominant - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the Grooved Pegboard test, non-dominant hand speed of completion (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 8 | 10 | 10
Z score | -0.16 (1.10) | -0.11 (0.53) | 0.20 (0.85) | 0.05 (0.85)

20. Secondary Outcome: Neurocognitive Performance: Grooved Pegboard, Non-Dominant - Per Protocol
Description: as for outcome 19
Time Frame: 24 Weeks
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | -0.17 (1.39) | 0.13 (0.61) | 0.41 (0.94) | -0.42 (0.84)

21. Secondary Outcome: Neurocognitive Performance: CalCAP, Choice - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the CalCAP Choice test, mean reaction time (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 10 | 6 | 11 | 8
Z score | 0.152 (1.468) | -0.570 (1.348) | 0.871 (2.771) | -1.325 (1.779)

22. Secondary Outcome: Neurocognitive Performance: CalCAP, Choice - Per Protocol
Description: as for outcome 21
Time Frame: 24 Weeks
Population: Per protocol analysis: Includes participants who completed the study per protocol and with test data available at the Baseline and Week 24 visits.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 1 | 8 | 5
Z score | -0.440 (1.004) | -1.17 (NA) — Mean based on only 1 participant | 1.724 (2.711) | -0.554 (1.751)

23. Secondary Outcome: Neurocognitive Performance: CalCAP, Sequential - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by the CalCAP Sequential test, mean reaction time (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 10 | 6 | 11 | 8
Z score | 0.272 (0.781) | -0.025 (0.931) | 0.317 (1.534) | -0.530 (0.535)

24. Secondary Outcome: Neurocognitive Performance: CalCAP, Sequential - Per Protocol
Description: as for outcome 23
Time Frame: 24 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 1 | 8 | 5
Z score | 0.355 (0.886) | -0.11 (NA) — Mean based on only 1 participant. | 0.631 (1.464) | -0.394 (0.433)

25. Secondary Outcome: Neurocognitive Performance: Symbol-Digit Test - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by Symbol-Digit Test score, number correct in 120 seconds (Z scores).
Time Frame: 24 Weeks
Population: Includes all participants who completed the study with test data available (no data substitution) at the Baseline and Week 24 visits for Intention to Treat analysis.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 9 | 10 | 10
Z score | 0.494 (0.828) | 0.175 (1.183) | 0.050 (0.901) | -0.175 (0.677)

26. Secondary Outcome: Neurocognitive Performance: Symbol-Digit Test - Per Protocol
Description: as for outcome 25
Time Frame: 24 Weeks
Population: Per protocol analysis: Includes participants who completed the study per protocol and with test data available (no data substitution) at the Baseline and Week 24 visits.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | 0.354 (0.666) | -0.167 (1.010) | 0.275 (0.975) | -0.180 (0.903)

27. Secondary Outcome: Neurocognitive Performance: Timed Gait - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by Timed Gait, three-trial average time (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 10 | 7 | 8 | 8
Z score | -0.575 (1.038) | -0.425 (1.135) | 0.283 (0.869) | -0.148 (1.127)

28. Secondary Outcome: Neurocognitive Performance: Timed Gait - Per Protocol
Description: Baseline to Week 24 change in neurocognitive performance as measured by Timed Gait, three-trial average time (Z scores).
Time Frame: 24 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 5 | 5
Z score | -0.641 (1.141) | -0.170 (1.465) | 0.574 (0.833) | -0.584 (1.166)

29. Secondary Outcome: Neurocognitive Performance: NPZ-8 - Intent to Treat
Description: Baseline to Week 24 change in neurocognitive performance as measured by NPZ-8 scores calculated for all participants who completed the trial with measurable Baseline and Week 24 data for at least 6 of the 8 data points. The data points that comprise the NPZ-8 include timed gait, symbol-digit, grooved pegboard dominant and non-dominant, CalCAP Choice reaction time and Sequential reaction time, Trail-making Test A and B. The baseline to week 24 changes for each test were averaged to get each change in NPZ-8 score.
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10
Z score | 0.121 (0.538) | -0.165 (0.590) | 0.313 (0.628) | -0.191 (0.432)

30. Secondary Outcome: Neurocognitive Performance: NPZ-8 - Per Protocol
Description: as for outcome 29
Time Frame: 24 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 5
Z score | -0.005 (0.527) | -0.298 (0.290) | 0.575 (0.485) | -0.199 (0.192)

31. Secondary Outcome: Change in CES-D Score - Intent to Treat
Description: Functional assessment: Change in Center for Epidemiologic Studies Depression Scale (CES-D) score between baseline and week 24 for all participants for whom baseline and follow-up CES-D data are available (intent to treat analysis).
Time Frame: 24 Weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10
units on a scale | -1.182 (6.750) | 1.222 (13.321) | -1.182 (2.822) | 2.600 (8.618)

32. Secondary Outcome: Change in CES-D Score - Per Protocol
Description: Functional assessment: Change in Center for Epidemiologic Studies Depression Scale (CES-D) score between baseline and week 24 for all participants for whom baseline and follow-up CES-D data are available (per protocol).
Time Frame: 24 Weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine and Fluconazole | Fluconazole | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 3 | 8 | 5
units on a scale | 1.667 (3.327) | 6.000 (16.093) | -0.875 (3.182) | 8.800 (7.190)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 24 week clinical trial period for each subject, and if pertinent, during the follow-up period, which was at least 14 days and up to 60 days after discontinuation of the intervention. When applicable, some adverse event data were collected between the screening visit and baseline visit (e.g., safety data pertaining to the lumbar puncture procedure).
Description: Routine safety blood tests were performed at screening, baseline, week 4, week 12, and week 24 visits. A combination of open-ended questioning, medical chart review, and standard questionnaires was used to collect adverse event data at each of the visits. A study clinician performed standard neuro-medical physical exams at baseline, week 12, and week 24. If warranted, data collection occurred between visits, ad hoc, to track ongoing adverse events, as well as after stopping the intervention.
Arm/Group | Paroxetine and Fluconazole | Paroxetine | Fluconazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/11 | 3/11 | 3/11
Other Adverse Events (participants affected / at risk) | 11/12 | 10/11 | 10/11 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine and Fluconazole (N=12) | Paroxetine (N=11) | Fluconazole (N=11) | Placebo (N=11)
Surgery, knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Inpatient elective surgery followed by complications
Heroin abuse, relapse (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose, non-fasting, high (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 4 (DAIDS); hyperglycemia in the context of acute uncontrolled diabetes
Surgery, neck (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Elective surgery to treat cervical stenosis
Depression, acute (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 3 (DAIDS); Acute episode, resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine and Fluconazole (N=12) | Paroxetine (N=11) | Fluconazole (N=11) | Placebo (N=11)
Abdominal cramping or pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Generalized abdominal cramping or pain (non-focalized)
Absolute neutrophil count (ANC), low (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Blood test, grade 2 (DAIDS 2.0)
Acute bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Grade 2 (DAIDS 2.0); context of chronic obstructive pulmonary disease requiring visit to emergency department
Agitation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase (ALT), high (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 1 (1) — Blood test, grade 2 (DAIDS 2.0)
Aspartate aminotransferase (AST), high (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 — Blood test, grade 2 (DAIDS 2.0)
Alkaline phosphatase, high (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 — Blood test, grade 2 (DAIDS 2.0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 | 1 (1) | 1 (1)
Altered taste (General disorders) | 0 | 1 (1) | 1 (1) | 0
Automobile accident (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 — Passenger, visit to ED, back injury, discharged home
Back pain, generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 | 0
Bilirubin, total, high (Hepatobiliary disorders) | 0 | 2 (5) | 3 (4) | 1 (1) — Blood test, grade 2 or 3 (DAIDS 2.0)
Blood urea nitrogen (BUN), high (Metabolism and nutrition disorders) | 3 (5) | 0 | 1 (3) | 3 (6) — Blood test, range: 23-41 mg/dL
Blood urea nitrogen (BUN), low (Metabolism and nutrition disorders) | 1 (1) | 0 | 1 (1) | 1 (1) — Blood test, range: 5-6 mg/dL
Chlamydia, new infection/exposure (Infections and infestations) | 0 | 0 | 1 (1) | 0 — Treated for infection
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 — Grade 2 or 3 (DAIDS 2.0)
Creatinine, blood, high (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (3) — Blood test, grade 2 (DAIDS 2.0)
Cyst, subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Darkening of urine (General disorders) | 0 | 1 (1) | 0 | 1 (1)
Depressed mood (Psychiatric disorders) | 0 | 0 | 2 (2) | 0 — Self-reported
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (2) — Grade 2 (DAIDS 2.0)
Dizziness (General disorders) | 2 (2) | 0 | 0 | 0 — Self-reported, intermittent
Dry mouth (General disorders) | 3 (3) | 0 | 2 (2) | 0 — Self-reported
Fatigue (General disorders) | 1 (1) | 0 | 0 | 0 — Grade 2 (DAIDS 2.0)
Flank pain, unilateral (General disorders) | 0 | 0 | 1 (1) | 0 — Non-specific, self-limited
Gastroenteritis, foodborne illness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) — Self-reported
Glucose, blood, high (Endocrine disorders) | 0 | 0 | 3 (4) | 1 (1) — Blood test, non-fasting, grade 2 or 3 (DAIDS 2.0)
Glucose, blood, low (General disorders) | 0 | 0 | 1 (1) | 1 (1) — Blood test, non-fasting, grade 2 (DAIDS 2.0)
Headache, non-specific (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 — Intermittent, grade 2 (DAIDS 2.0)
Headache, post-lumbar puncture (Nervous system disorders) | 1 (1) | 0 | 0 | 1 (1) — Post-LP postural headache requiring follow-up care
Hypokalemia (General disorders) | 1 (2) | 0 | 0 | 0 — Grade 2 (DAIDS 2.0)
Incontinence, acute nocturnal (General disorders) | 0 | 0 | 1 (1) | 0 — Self-limited
Insomnia (General disorders) | 0 | 2 (2) | 1 (1) | 0
Joint pain, generalized (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (1) | 0
Joint pain, hip, unilateral (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0
Joint pain, shoulder, unilateral (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0
Lightheadedness (General disorders) | 1 (1) | 0 | 1 (1) | 0
Lymph node infection, neck (Infections and infestations) | 0 | 0 | 1 (1) | 0 — Treated for infection
Lymphadenopathy, cervical (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4) | 1 (1) — Grade 2 or 3 (DAIDS 2.0)
Nephrolithiasis (kidney stone) (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertensive episode (Cardiac disorders) | 0 | 0 | 0 | 1 (1) — Grade 3 (DAIDS); context of diagnosed/treated hypertension, participant had not taken morning medications
Nose bleed (General disorders) | 0 | 0 | 1 (1) | 0 — Self-limited
Polyuria (General disorders) | 1 (1) | 0 | 0 | 0 — Self-limited
Prostitis (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0
Psychotropic effects, non-specific (General disorders) | 0 | 1 (1) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 4 (4) | 1 (1) | 0
Sprain, ankle (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Syphilis, new infection/exposure (Infections and infestations) | 1 (1) | 0 | 1 (1) | 0 — Treated for infection
Tinnitus, bilateral (General disorders) | 0 | 1 (1) | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 — Treated for infection
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary hesitancy (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0
Visual changes (Eye disorders) | 0 | 0 | 1 (1) | 0
Vivid or disturbing dreams (General disorders) | 0 | 2 (2) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 — Grade 2 (DAIDS 2.0)
Weight loss (General disorders) | 0 | 0 | 1 (1) | 0 — Grade 2 (DAIDS 2.0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes